CLINICAL TRIAL: NCT04497584
Title: An Investigator-sponsored Phase 2 Trial of Afatinib Plus Prednisone for Advanced Squamous Non-small Cell Lung Cancer
Brief Title: Phase 2 Trial of Afatinib Plus Prednisone for Advanced Squamous NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sheena Bhalla, Assistant Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2020-1363
Record Dates: First submitted 2020-05-22; First posted 2020-08-04 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — Afatinib; Prednisone

STUDY DESIGN:
Intervention Model Description: Afatinib 40 mg PO daily Prednisone 40 mg PO daily (starting 7 days after afatinib)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Afatinib + Prednisone (Experimental): Afatinib 40 mg PO daily
  Prednisone 40 mg PO daily starting 7 days after Afatinib
  Interventions: Drug: Afatinib + Prednisone

INTERVENTIONS:
Drug: Afatinib + Prednisone — Afatinib (40mg) will be taken by mouth daily starting on Cycle 1, Day -7. Prednisone (40mg) will be taken by mouth daily starting on Cycle 1, Day 1.

SUMMARY:
To determine the efficacy of combined afatinib and prednisone in previously treated advanced squamous NSCLC

DETAILED DESCRIPTION:
This two-stage phase 2 study will determine the safety, tolerability, recommended phase 2 dose/maximum tolerated dose, preliminary efficacy and predictive/pharmacodynamic biomarkers of combined EGFR inhibition (afatinib) and TNF inhibition (prednisone) in previously treated NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure.
* Previously treated (up to three prior lines of therapy), histologically proven advanced squamous NSCLC.
* No prior treatment with EGFR inhibitors, IMIDs (eg, thalidomide, lenalidomide), or anti-TNF antibodies.
* No treatment with systemic glucocorticoids within 3 weeks of initiation of study therapy (topical and inhaled glucocorticoids are permitted).
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ and marrow function as defined below:
* absolute neutrophil count ≥ 1,000/μL
* platelets ≥ 50,000/μl
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
* CrCl ≥ 45 ml/min
* For both male and female patients, effective methods of contraception must be used throughout the study and for 3 months following the last dose of study treatment.
* Adequate archival tissue (5-10 slides) for correlative studies.
* Subject must have measurable disease per RECIST 1.1

Exclusion Criteria:

* Chemotherapy, radiotherapy, or other cancer therapy within two weeks prior to starting study treatment. Subjects must have recovered from prior treatment-related to toxicities to grade 1 or baseline (excluding alopecia and clinically stable toxicities requiring ongoing medical management, such as hypothyroidism from prior immune checkpoint inhibitor treatment).
* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* Symptomatic brain metastases or brain metastases requiring escalating doses of corticosteroids
* History of hypersensitivity or allergic reactions attributed to afatinib or prednisone.
* Uncontrolled intercurrent illness including but not limited to poorly controlled diabetes (which may worsen in setting of chronic prednisone therapy), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival of combined afatinib and prednisone in previously treated NSCLC | From date of enrollment to date of documented progression or death from any cause, whichever came first, assessed up to 60 months
  Measure progression-free survival rate.

SECONDARY OUTCOMES:
Response rate of combined afatinib and prednisone in previously treated NSCLC | From date of enrollment to date of documented progression or death from any cause, whichever came first, assessed up to 60 months
  Measure response rate by evaluation of target lesions by measuring disease.
Overall survival of combined afatinib and prednisone in previously treated NSCLC | From date of enrollment to date of documented progression or death from any cause, whichever came first, assessed up to 60 months
  Measure Overall Survival, as the time from the date of initiation of study treatment until death of any cause.
Safety of combined afatinib and prednisone in previously treated NSCLC | From date of enrollment to date of documented progression or death from any cause, whichever came first, assessed up to 60 months
  Measure risk to study participants by completing blood test and assessing according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sheena Bhalla, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No